CLINICAL TRIAL: NCT03909607
Title: Comparison of Nebulized Sub-dissociative Dose Ketamine at Three Different Dosing Regimens for Treating Acute and Chronic Painful Conditions in the ED: A Prospective, Randomized Trial
Brief Title: Nebulized Sub-dissociative Dose Ketamine for Treating Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager; co-investigator, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-11-12
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SDK 0.75 mg/kg (Active Comparator): The patients will receive sub-dissociative ketamine at a dose of 0.75mg/k
  Interventions: Drug: Ketamine 0.75 mg/kg
- SDK 1.0 mg/kg (Active Comparator): The patients will receive sub-dissociative ketamine at a dose of 1.0mg/k
  Interventions: Drug: Ketamine 1.0 mg/kg
- SDK 1.5 mg/kg (Active Comparator): The patients will receive sub-dissociative ketamine at a dose of 1.5mg/k
  Interventions: Drug: Ketamine 1.5 mg/kg

INTERVENTIONS:
Drug: Ketamine 0.75 mg/kg — Patients with moderate to severe pain will receive Ketamine at a dose of 0.75mg/kg
  Arms: SDK 0.75 mg/kg
Drug: Ketamine 1.0 mg/kg — Patients with moderate to severe pain will receive Ketamine at a dose of 1.0 mg/kg
  Arms: SDK 1.0 mg/kg
Drug: Ketamine 1.5 mg/kg — Patients with moderate to severe pain will receive Ketamine at a dose of 1.5 mg/kg
  Arms: SDK 1.5 mg/kg

SUMMARY:
The investigators previous research study comparing the efficacy of intravenous ketamine to morphine showed ketamine to provide equivalent relief of moderate to severe acute pain in emergency department patients. A second study by the investigators showed that increasing the time of administration of the ketamine, from a push injection to a drip infusion, will minimize the adverse effects experienced by recipients of ketamine.

The investigators now aim to see if nebulized subdissociative-dose ketamine administered as a single agent in a dose of 1.5 mg/kg via Breath-Actuated Nebulizers (BAN) over 5-15 minutes will provide a better pain relief in comparison to 1 mg/kg and 0.75 mg/kg doses or if the lower doses are equally as effective.

DETAILED DESCRIPTION:
STUDY DESIGN

Subjects: Patients 18 years of age and older presenting to the ED with acute and chronic painful conditions such as traumatic and non-traumatic abdominal, flank, back, or musculoskeletal pain as well as exacerbation of chronic abdominal, musculoskeletal and neuropathic pain with a score of 5 or more on a standard 11- point (0 to 10) numeric rating scale and requiring sub-dissociative dose ketamine analgesia, as determined by the treating attending physician. Patients' screening and enrollment will be performed by study investigators and research assistants. All patients will be enrolled at various times of the day when study investigators will be available for patient enrollment and an ED pharmacist will be available for medication preparation

Eligibility Criteria: Patients 18 years of age and older presenting to the ED with acute and chronic painful conditions such as traumatic and non-traumatic abdominal, flank, back, or musculoskeletal pain as well as exacerbation of chronic abdominal, musculoskeletal and neuropathic pain with a score of 5 or more on a standard 11- point (0 to 10) numeric rating scale.

Exclusion Criteria: Altered mental status, allergy to ketamine, pregnant patients, weight greater than 150 kg, unstable vital signs (systolic blood pressure <90 or>180 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min), inability to provide consent, and past medical history of alcohol or drug abuse, or schizophrenia.

Design: This is a prospective, randomized, double-blind trial comparing analgesic efficacy and safety of nebulized SDK administered at three different doses to patients presenting to the ED of Maimonides Medical Center with acute and chronic painful conditions. Upon meeting the eligibility criteria, patients will be randomized into one of three study arms based on the dosing of the SDK: 0.75 mg/kg, 1 mg/kg, and 1.5 mg/kg.

Data Collection Procedures: Each patient will be approached by a study investigator for acquisition of written informed consent and Health Insurance Portability and Accountability Act authorization after being evaluated by the treating emergency physician and determined to meet study eligibility criteria. When English will not be the participant's primary language, a staff interpreter or licensed telephone interpreter would be used. Baseline pain score will be determined with an 11-point numeric rating scale (0 to 10), described to the patient as "no pain" being 0 and "the worst pain imaginable" being 10. A study investigator will record the patient's body weight and baseline vital signs. The on-duty ED pharmacist will prepare a breath-actuated nebulizer with doses of 0.75 mg/kg, 1 mg/kg, and 1.5 mg/kg according to the predetermined randomization list, which will be created in SPSS (version 24; IBM Corp, Armonk, NY) with block randomization of every 10 participants. The medication will be delivered to the treating nurse in a blinded fashion and will be administered via breath-initiated nebulization with a minimum time of 5 min and maximum time of 15 min up to three doses.

Study investigators will record pain scores, vital signs, and adverse effects at 15, 30, 60, 90, and 120 minutes. If patients reported a pain numeric rating scale score of 5 or greater and requested additional pain relief, a second (equivalent to the first dose) of SDK via BAN will be administered to the patient in a blinded fashion. In situations when nebulized SDK will fail to achieve acceptable (by patient) pain relief or patient will refuse to continue nebulized SDK treatment, morphine at 0.1 mg/kg will be administered as a rescue analgesic.

All data will be recorded on data collection sheets, including patients' sex, demographics, medical history, and vital signs and entered into SPSS (version 24.0; IBM Corp) by the research manager. Development of the randomization list, confirmation of written consent acquisition for all participants, and statistical analyses will be conducted by the research manager and statistician, who would work independent of any data collection.

Patients will be closely monitored for any change in vital sings and for adverse effects during the entire study period (up to 2 h) by study investigators. Common adverse effects that are associated with sub-dissociative dose ketamine are felling of unreality, dizziness, nausea, vomiting, and sedation.

Data Analysis: Data analyses will include frequency distributions, paired t-test to assess a difference in pain scores within each group, and independent-sample t-test to assess differences in pain scores between the 3 groups at the various intervals.

Mixed-model linear regression will be used to compare changes in pain numeric rating scale across time points. This will compensate for participants lost to follow-up and allow all patients' data to be analyzed on an intention-to-treat principle.

For categorical outcomes (eg, complete resolution of pain), a X2 or Fisher's exact test will be used to compare outcomes at 30 minutes. Percentage differences and 95% confidence intervals between the treatment groups will be calculated for all time points with P<.05 to denote statistical significance. Based on the validation of a verbally administered rating scale of acute pain in the ED and the comparison of verbal and visual pain scales, we will use a primary outcome consisting of a minimal clinically meaningful difference of 1.3 between three groups at the 30-minute pain assessment.28,29

Sample Size: Assuming an SD of 3.0, a power analysis determined that a repeated-measures ANOVA with a sample size of 34 patients per group ( 102 total) will provide at least 80% power to detect a difference of at least 1.3 at 30 minutes (as well as at any other interval post-baseline), with an alpha=.05. To account for possible missing data the total sample size will be 120 patients (40 per group).A pre-planned interim data analysis will occur upon reaching a total of total of 60 patients ( 20) patients per group.

Expected Outcomes: The primary outcome will include a comparative reduction of pain scores on numeric rating pain scale (NRS) between recipients of nebulized SDK at three different doses at 30 minutes post-analgesic administration. The secondary outcomes will include a need for second or third dose, a need for rescue analgesia at either 30 or 60 minutes and adverse events in each group. With respect to unique adverse effects of SDK, we will use Side Effect Rating Scale for Dissociative Anesthetics (SERSDA) and Richmond Agitation Sedation Scale (RASS) (ref) SERSDA Scale includes fatigue, dizziness, nausea, headache, feeling of unreality, changes in hearing, mood change, general discomfort, and hallucinations with severity of each graded by patients on a five-point scale, with "0" representing the absence of any adverse effects and "4" representing a severely bothersome side effect. RASS evaluates the severity of agitation and/or sedation in accordance to the nine-point scale with scores ranging from "-4" (deeply sedated) to "0" (alert and calm) to "+4" (combative).

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* acute and chronic abdominal, flank, back, musculoskeletal pain, and traumatic pain as well as cancer pain
* initial pain score of 5 or more on a standard 11- point (0 to 10) numeric rating scale.

Exclusion Criteria:

* altered mental status,
* allergy to ketamine,
* weight greater than 150 kg,
* unstable vital signs (systolic blood pressure <90 or>180 mm Hg,
* pulse rate <50 or >150 beats/min,
* respiration rate <10 or >30 breaths/min)
* alcohol or drug abuse
* inability to provide consent
* psychiatric illness (schizophrenia),
* recent (4 hours before) opioid use.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SDK 0.75 mg/kg | SDK 1.0 mg/kg | SDK 1.5 mg/kg
Started | 40 | 40 | 40
Completed | 35 | 36 | 38
Not Completed | 5 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SDK 0.75 mg/kg | SDK 1.0 mg/kg | SDK 1.5 mg/kg | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (20) | 51 (16) | 50 (18) | 51 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 23 | 68
  Male | 17 | 18 | 17 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 40 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores From Baseline to 30 Minutes
Description: Patients will be assessed via an 11 point Likert numeric rating scale at time medication is given (baseline) and 30 minutes later. The difference in pain scores will be assessed between the 3 groups. The numeric rating scale range is from 0 to 10 with 0 being no pain and 10 being very severe pain.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SDK 0.75 mg/kg | SDK 1.0 mg/kg | SDK 1.5 mg/kg
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 4.0 (1.9) | 4.2 (2.1) | 4.1 (1.9)

ADVERSE EVENTS:
Time Frame: 120 minutes
Arm/Group | SDK 0.75 mg/kg | SDK 1.0 mg/kg | SDK 1.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 5/40 | 14/40 | 15/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SDK 0.75 mg/kg (N=40) | SDK 1.0 mg/kg (N=40) | SDK 1.5 mg/kg (N=40)
Dizzines (Nervous system disorders) | 5 (5) | 14 (14) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT03909607/Prot_SAP_000.pdf